CLINICAL TRIAL: NCT03696381
Title: Clinical Trial of The Boosting Effect of Transcranial Random Noise Stimulation (tRNS) in Cognitive Rehabilitation of Patients With Traumatic Brain Injury
Acronym: TRUST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Guttmann (Other)
Responsible Party: Principal Investigator, Adria Garcia Rosas, PhD Student, Institut Guttmann
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-281
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Traumatic Brain Injury; Cognitive Impairment
Keywords: computerized cognitive rehabilitation; trns; traumatic brain injury; tbi; cognitive impairment
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tRNS (Experimental): Real tRNS + Guttmann NeuroPersonalTrainer (GNPT) 3 days per week over 8 weeks.
  Interventions: Other: Real tRNS
- Sham tRNS (Sham Comparator): Sham tRNS + Guttmann NeuroPersonalTrainer (GNPT) 3 days per week over 8 weeks.
  Interventions: Other: Sham tRNS

INTERVENTIONS:
Other: Real tRNS — The treatment consists of a set of 1-h sessions, three sessions per week for 8 weeks. A series of cognitive exercises of attention, memory, and executive functions will be conducted in each session. During the first 20 minutes of each cognitive training session, patients will receive bi-frontal and bi-parietal tRNS. It has a start and end ramp of two seconds in each case to avoid the slight unpleasant sensation that occurs in the first moments of the introduction of direct current DC.
  Other Names: Guttmann, NeuroPersonalTrainer (GNPT)
  Arms: Real tRNS
Other: Sham tRNS — The treatment consists of a set of 1-h sessions, three sessions per week for 8 weeks. A series of cognitive exercises of attention, memory, and executive functions will be conducted in each session. We will apply a sham tRNS for the first 20 minutes of each cognitive training session. The subjects will receive sham tRNS and will perform the same type of cognitive training as the rest of patients and will receive the same type of adverse reaction questionnaire. Subjects receiving simulated stimulation will receive the same type of ramps at the beginning and end of the session to ensure triple-blind maintenance .
  Other Names: Guttmann, NeuroPersonalTrainer (GNPT)
  Arms: Sham tRNS

SUMMARY:
The main objective of this study is to evaluate the effects of tRNS while undergoing computerized cognitive rehabilitation therapy to conclude if this combination of therapies would be effective for the cognitive rehabilitation of patients with acquired brain damage, such as traumatic brain injury. We want to study the therapeutic potential of tRNS to enhance the therapeutic outcome of cognitive training, studying its global effect over the rehabilitation of attention, memory and executive functions, compared to sham tRNS.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* documented history of severe or moderate TBI (severe TBI: Glasgow Coma Scale 3-8; moderate TBI: Glasgow Coma Scale 9-13)
* out of post-traumatic amnesia
* less than 6 months after TBI
* cognitive impairment objectified by neuropsychological exploration.

Exclusion Criteria:

* impairment of language, affecting the production and/or comprehension of speech and the ability to read and/or write
* severe alteration of the visual field or visual perception problems that limits the use of technological devices
* sever motor impairment of both upper extremities that prevent the use of technological devices
* previous or current history of psychiatric, neurological or systemic alterations that affect the central nervous system
* history of substance abuse
* dermatological diseases in the skull
* presence of metal implants or holes in the skull
* epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Conners Continuous Performance Test (CPT-II) | 1 day
  To improve performance in sustained attention after receiving experimental intervention.
Digit Span Forward from the Wechsler Adult Intelligence Scale | 1 day
  To improve performance in span of immediate verbal recall after receiving experimental intervention.
Digit Span Backward from the Wechsler Adult Intelligence Scale | 1 day
  To improve performance in working memory after receiving experimental intervention.
Rey Auditory Verbal Learning Test | 1 day
  To improve performance in short-term, long-term and recognition.
Letters and Numbers from the Wechsler Adult Intelligence Scale | 1 day
  To improve performance in working memory after receiving experimental intervention.
Spanish phonemic fluency test (PMR) | 1 day
  To improve performance in phonemic fluency after receiving experimental intervention.

SECONDARY OUTCOMES:
Trail Making Test A (TMT-A) | 1 day
  To improve performance in visual attention
Trail Making Test B (TMT-B) | 1 day
  To improve performance in task-switching
Wisconsin Card Sorting Test (WCST) | 1 day
  To improve performance in set-shifting
Stroop Color and Word test (Stroop Test) | 1 day
  To improve performance in inhibitory control

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain